CLINICAL TRIAL: NCT02627417
Title: Prospective Multicenter Randomized Open-label Controlled Trial Assessing Efficacy and Safety of DAPSone as a Second-line Option in Adult Immune Thrombocytopenia
Brief Title: Efficacy and Safety of DAPSone as a Second-line Option in Adult Immune Thrombocytopenia
Acronym: DAPS-ITP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P140925
Record Dates: First submitted 2015-11-03; First posted 2015-12-11 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Adult Immune Thrombocytopenia (ITP); Dapsone
Keywords: ITP; Dapsone
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Dapsone; Prednisone; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dapsone: (Disulone®) (Experimental): Dapsone: Disulone® given orally at 100 mg per day
  Interventions: Drug: Dapsone (Disulone®); Drug: Prednisone (Cortancyl®)
- Prednisone (Cortancyl®) alone and "standard of care" (Active Comparator): Prednisone (Cortancyl®) alone at 1 mg/kg for 3 weeks followed by monitoring and "standard of care" (control arm)
  Interventions: Drug: Prednisone (Cortancyl®) alone followed by monitoring and "standard of care"

INTERVENTIONS:
Drug: Dapsone (Disulone®) — Experimental group will receive dapsone at a fixed dose of 100 mg per day for a total of 12 months unless they fail to respond to the treatment.
  Other Names: experimental arm
  Arms: Dapsone: (Disulone®)
Drug: Prednisone (Cortancyl®) alone followed by monitoring and "standard of care" — Patients randomized in the control arm will be treated only prednisone at a daily dose of 1 mg per kg for 2 weeks and then tapered and stopped over a week for a total of 3 consecutive weeks. After this 3 weeks period, patients from arm B will be left without treatment and monitored.
  Other Names: control arm
  Arms: Prednisone (Cortancyl®) alone and "standard of care"
Drug: Prednisone (Cortancyl®) — Experimental group will receive prednisone at a daily dose of 1 mg per kg for 2 weeks and then tapered and stopped over a week for a total of 3 consecutive weeks.
  Other Names: experimental arm
  Arms: Dapsone: (Disulone®)

SUMMARY:
Due to its expected efficacy based on the retrospective data available in ITP, its relatively good safety profile and its very low cost , dapsone could be a good steroid-sparing second-line option for adults with ITP.

This study is a phase III prospective multicenter randomized open trial comparing two treatment strategies:

* Arm A (experimental arm): prednisone at 1 mg/kg for 3 weeks + dapsone at 100 mg per day up to week 52 if an initial response is achieved.
* Arm B (control arm): prednisone alone at 1 mg/kg for 3 weeks followed by monitoring and "standard of care" The aim of the study is to demonstrate the efficacy of dapsone based on the overall response rate (including response and complete response) as a second-line treatment for adults with newly-diagnosed persistent or chronic (modified by amendment 08/11/2016) ITP not achieving a durable response with corticosteroids. The primary endpoint will be the overall response-rate (response or complete response according to standard definitions) in both arms at week 52 (1 year).

The secondary endpoints are the following :

* To assess the safety of dapsone over the study period and especially the incidence of cutaneous reactions.
* To analyze the overall response rate (platelet count > 30 x 109/L with at least a doubling of the pre-treatment count in the absence of any other ITP treatment) in both treatment arms at week 24.
* To compare the rate of complete response and failure in both arms at 24 and 52 weeks.
* To compare time to treatment failure (TTF) in both arms
* To investigate the mechanisms of action of dapsone in ITP in a subgroup of patients (ancillary study)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of primary ITP according to the standard definition and international guidelines.
* Previous transient response to corticosteroids ± intravenous immunoglobulin defined by an increase of the platelet count above 30 x 109/L with at least a twofold increase of the pre-treatment count.
* At least platelet count ≤ 30 x 109/L within the 2 weeks before inclusion with a platelet count at time of inclusion below 50 x 109/L, or platelet count < 50 x 109/L at any time point in patients requiring treatment (i.e., patients with bleeding symptoms, elderly patients with comorbidities and/or patients on aspirin for example, or other reason at the investigator discretion) (modified by amendment 8/11/2016)
* Normal marrow aspirate for patients aged of 60 and above.
* Negative pregnancy test and effective method of contraception for women of childbearing age over the study period.
* Informed consent.
* Patient affiliated to the French National Social Security System

Exclusion Criteria:

* Secondary ITP. Patients with positive antinuclear antibodies and/or positive antiphospholipid antibodies not fulfilling the classification criteria for systemic lupus erythematosus and/or antiphospholipid antibody syndrome will not be excluded.
* Platelet count ≥ 50 x 109/L or between 30 and 50 x 109/L and no bleeding symptoms and no need for treatment (modified by amendment 8/11/2016)
* Severe bleeding manifestations defined a bleeding score ≥ 8
* No previous transient response to corticosteroids ± intravenous immunoglobulin.
* Previous ITP treatment other than corticosteroids and intravenous immunoglobulin (including rituximab and splenectomy).
* Active severe infection or history of severe infection within 4 weeks before inclusion.
* History of allergy to sulfonamides.
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency.
* History of methemoglobinemia
* Hemoglobin level < 11g/dL and/or neutrophil count < 1,500/ gL.
* History of autoimmune (Evans' syndrome) or hereditary haemolytic anemia.
* Liver or kidney function impairment (creatinine clearance < 30 ml/min, ALT, AST >2 times upper normal limit). (modified by amendment 8/11/2017)
* Hepatitis C virus (HCV) Ab, HIV Ab, HBsAg, seropositive status. (modified by amendment 8/11/2017)
* Concomitant medical condition requiring anticoagulation. (modified by amendment 8/11/2017)
* Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2015-12; Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Overall response-rate. | at week 52

SECONDARY OUTCOMES:
Assess the safety of dapsone especially the incidence of cutaneous adverse effects. | over the study period (up to 52 weeks)
Compare the overall response rate . | at week 24
  platelet count > 30 x 109/L with at least a doubling of the pre-treatment count in the absence of any other ITP treatment in both arms
Proportion of patients with complete response in both arms, defined as follows: - Proportion of patients with a platelet count > 100 x 109/L in the absence use of any other ITP directed therapies | at 24 and at 52 weeks
Proportion of non-responders patients (primary failure) | at 24 and at 52 weeks
  Patients will be considered as being non-responders if:
  1. Their platelet count at the end of the study is < 30 x 109/L, but also, in the setting of this study if:
  2. They need a rescue therapy (a new course of corticosteroids and/or intravenous immunoglobulin) more than 6 weeks after inclusion.
     or
  3. They receive any other treatment for ITP than dapsone or prednisone (including rituximab, splenectomy and Tpo-R agonists) over the study period
Number of days to treatment failure in both arms | over the study period (up to 52 weeks)
Mechanisms of action of Dapsone: degree of phagocytosis of autologous platelets and red blood cells, cytokines profile expression (including IL-8), whole blood gene expression signature between responders and non-responders. | over the study period (52 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: MARC MICHEL, Prof. M.D, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France

REFERENCES:
- [Background] Durand JM, Lefevre P, Hovette P, Mongin M, Soubeyrand J. Dapsone for idiopathic autoimmune thrombocytopenic purpura in elderly patients. Br J Haematol. 1991 Jul;78(3):459-60. doi: 10.1111/j.1365-2141.1991.tb04467.x. No abstract available. PMID 1873232
- [Background] Godeau B, Oksenhendler E, Bierling P. Dapsone for autoimmune thrombocytopenic purpura. Am J Hematol. 1993 Sep;44(1):70-2. doi: 10.1002/ajh.2830440117. PMID 8342569
- [Background] Hernandez F, Linares M, Colomina P, Pastor E, Cervero A, Perez A, Perella M. Dapsone for refractory chronic idiopathic thrombocytopenic purpura. Br J Haematol. 1995 Jun;90(2):473-5. doi: 10.1111/j.1365-2141.1995.tb05179.x. PMID 7794776
- [Background] Godeau B, Durand JM, Roudot-Thoraval F, Tenneze A, Oksenhendler E, Kaplanski G, Schaeffer A, Bierling P. Dapsone for chronic autoimmune thrombocytopenic purpura: a report of 66 cases. Br J Haematol. 1997 May;97(2):336-9. doi: 10.1046/j.1365-2141.1997.412687.x. PMID 9163598
- [Background] Damodar S, Viswabandya A, George B, Mathews V, Chandy M, Srivastava A. Dapsone for chronic idiopathic thrombocytopenic purpura in children and adults--a report on 90 patients. Eur J Haematol. 2005 Oct;75(4):328-31. doi: 10.1111/j.1600-0609.2005.00545.x. PMID 16146539
- [Derived] Larue M, Moulis G, Rueter M, Audia S, Comont T, Terriou L, Viallard JF, Pan-Petesch B, Royer B, Bonnotte B, Galicier L, Lambotte O, Lefrere F, Cheze S, Ebbo M, Duong TA, Boutin E, Languille L, Mahevas M, Godeau B, Canoui-Poitrine F, Michel M. Efficacy and safety of dapsone in adult primary immune thrombocytopenia. Blood Adv. 2025 Apr 22;9(8):1976-1983. doi: 10.1182/bloodadvances.2024014939. PMID 39874521